CLINICAL TRIAL: NCT05629702
Title: A Randomised Controlled Phase II Trial of Temozolomide With or Without Cannabinoids in Patients With Recurrent Glioblastoma
Brief Title: ARISTOCRAT: Blinded Trial of Temozolomide +/- Cannabinoids
Acronym: ARISTOCRAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University of Leeds (Other); The Brain Tumour Charity (Other); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RG_21-001; 2021-005214-34 (EudraCT Number); ISRCTN (Registry Identifier: ISRCTN11460478)
Record Dates: First submitted 2022-11-07; First posted 2022-11-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Brain Tumor; Cannabis; Brain Tumor, Recurrent
Keywords: cannabinoid; GBM; temozolomide; sativex; nabiximols; cannabis; glioblastoma; brain; recurrent
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Marijuana Abuse; Recurrence | interventions — nabiximols; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Temozolomide with Nabiximols (Experimental): * Temozolomide 150mg/m2 for cycle 1, increasing to 200mg/m2 for subsequent cycles, once daily for days 1-5, orally, at the start of each 28 day cycle, up to a maximum of 6 cycles.
  * Nabiximols up to 12 oromucosal sprays per day up to a maximum of 6 cycles; self titrated over days 1-14 in cycle 1.
  Interventions: Drug: Nabiximols; Drug: Temozolomide
- Standard Temozolomide with Nabiximols-matched placebo (Placebo Comparator): * Temozolomide 150mg/m2 for cycle 1, increasing to 200mg/m2 for subsequent cycles, once daily for days 1-5, orally, at the start of each 28 day cycle, up to a maximum of 6 cycles.
  * Nabiximols-matched placebo up to 12 oromucosal sprays per day up to a maximum of 6 cycles; self titrated over days 1-14 in cycle 1.
  Interventions: Drug: Temozolomide; Drug: Nabiximols-matched placebo

INTERVENTIONS:
Drug: Nabiximols — Oromucosal spray
  Other Names: Sativex
  Arms: Standard Temozolomide with Nabiximols
Drug: Temozolomide — Oral capsule
Drug: Nabiximols-matched placebo — Nabiximols-matched placebo oromucosal spray
  Arms: Standard Temozolomide with Nabiximols-matched placebo

SUMMARY:
ARISTOCRAT is a phase II, multi-centre, double-blind, placebo-controlled, randomised trial to compare the cannabinoid Nabiximols with placebo in patients with recurrent MGMT methylated glioblastoma (GBM) treated with temozolomide (TMZ).

DETAILED DESCRIPTION:
This is a phase II, multi-centre, double-blind, placebo-controlled, randomised trial to compare the cannabinoid Nabiximols (Sativex®) with placebo in patients with recurrent MGMT methylated glioblastoma treated with temozolomide (TMZ). The trial will randomise a target number of 120 patients on a 2:1 basis to receive either Nabiximols or Nabiximols-matched placebo, in combination with standard TMZ.

Patients will be followed up at 4-weekly assessments for a minimum of 52 weeks from the start of trial treatment or until death, whichever is sooner. MRI scanning will be performed at screening, week 10, week 22, week 30, then 3-monthly after commencing trial treatment as per standard practice.

The trial includes an initial feasibility study of 40 patients to confirm safety, compliance and achievability of planned target recruitment. There are no formal criteria for evaluation of feasibility but once 40 patients have been recruited, the independent Data Monitoring Committee will review the adverse event data, details on protocol treatment received, monthly recruitment rates and projected recruitment in order to make recommendations on trial continuation.

The original phase II trial design allowed potential expansion of recruitment into a phase III trial, should the emerging phase II results warrant this development; however, the trial was revised to a standard phase II design to lower the recruitment targets in 2025

The trial will be linked to the Tessa Jowell BRAIN MATRIX (TJBM) programme; utilising TJBM infrastructure, opening the same participating sites, and aligning the data collection and Quality of Life assessments already embedded in TJBM. This collaboration will allow data sharing within the platform thereby streamlining patient entry and provide additional oversight through TJBM. Patients recruited to TJBM who are potentially eligible for ARISTOCRAT may be identified and suggested to sites for consideration to the trial.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of MGMT promoter methylated, IDH wild type (WT) GBM with consistent local molecular pathology (repeat biopsy at recurrence is NOT required).
* First recurrence of GBM planned for systemic treatment as determined by local Multidisciplinary Team (MDT), including agreement of a Consultant Neuro-Radiologist that imaging changes are most in keeping with recurrence and not pseudo-progression. Patients with a prior recurrence treated by surgical resection alone are eligible at time of first recurrence planned for systemic treatment.
* Patients must have received initial first-line treatment with standard dose conventionally fractionated radiotherapy (i.e. 40 Gy in 15 fractions or 54-60 Gy in 28-33 fractions; other regimes may be considered in consultation with the ARISTOCRAT Trial Office) with concomitant and adjuvant TMZ.

  * A minimum of 3 cycles of adjuvant TMZ must have been received.
  * A minimum of Stable Disease (SD) (or Partial Response (PR)/Complete Response (CR)) at the end of first-line treatment (measured by Response Assessment for Neuro-Oncology (RANO) criteria).
* ≥3 months since day 28 of the last cycle of TMZ.
* Karnofsky Performance Status ≥60.
* Adequate hematologic, renal, and hepatic function within 14 days prior to randomisation:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L
  * Platelet count ≥100 x 109/L
  * Serum creatinine clearance (measured or calculated (using local standard practice)) >30ml/min
  * Total serum bilirubin ≤1.5 x upper limit of normal (ULN)
  * Liver transaminases <2.5 x ULN
* If surgery has been performed for first recurrence, then the wound must be adequately healed and there must be residual enhancing disease on MRI within 21 days of surgery or new enhancement at later follow up deemed suitable for systemic treatment.
* Recovered from previous treatment side-effects ≤ Grade 2.
* If on systemic steroids, must be on stable (≥7 days) or decreasing dose of steroids.
* Willing and able to provide trial-specific informed consent.
* Willing and able to comply with trial requirements.
* Age ≥16.
* Able to start treatment within 28 days of randomisation.

Exclusion Criteria:

* Pathology inconsistent with IDH WT GBM (e.g. patients with molecular features of PXA or BRAF mutation will be excluded).
* Prior invasive malignancy (except non-melanoma skin cancer), unless disease free for a minimum of one year.
* Prior treatment with stereotactic radiotherapy, brachytherapy or Convection Enhanced Delivery (CED) of any agent.
* Prior treatment, apart from debulking surgery, for first recurrence of GBM.
* Any active co-morbidity making patient unsuitable for trial treatment in the view of the Investigator.
* Personal history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric diagnosis other than depression associated with their underlying glioma condition.
* Prior allergic reaction or significant toxicity (≥Grade 3 CTCAE) related to TMZ treatment.
* Current or recent cannabis or cannabinoid-based medications within 28 days of randomisation and/or unwilling to abstain for the duration of the trial.
* Women who are pregnant, breastfeeding or a woman of childbearing potential who is unwilling to use effective contraceptive methods during trial treatment and for 6 months after completion of trial treatment.

  o Women of childbearing age must have a negative pregnancy test within 7 days prior to randomisation.
* Men who are sexually active and unwilling/unable to use medically acceptable forms of contraception during trial treatment or for 6 months after completion of trial treatment.
* Contra-indication to MRI or gadolinium.
* Hereditary galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Known hypersensitivity to cannabinoids or excipients of the IMP.
* Known history of current or prior alcohol or drug dependence.
* Known Hepatitis B (HBV), Cytomegalovirus (CMV) or opportunistic infection.
* Has received a live vaccine within 28 days prior to randomisation.
* Unable to administer oromucosal medication due to mucosal lesions or other issues.
* Participation in another therapeutic clinical trial whilst taking part in this trial.
* Any psychological, familial, sociological or geographical condition hampering protocol compliance.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival time (OS) | Time in whole days from date of randomisation to the date of death from any cause, assessed at a minimum of 12 months..
  To establish whether the addition of cannabinoids (Nabiximols) to standard TMZ treatment improves overall survival time (OS) in MGMT methylated recurrent GBM compared to the addition of placebo to TMZ.

SECONDARY OUTCOMES:
Overall survival at 12 months (OS12) (and 6 and 24 months) | 6, 12 and 24 months
  Of particular clinical relevance is the overall survival at 12 months from date of randomisation, i.e. whether the participant is alive or not at that time point. Overall survival at 6 months and 24 months will also be of interest.
Progression-free survival time (PFS) | Time in whole days from the date of randomisation to the date of the first documented evidence of disease progression or death (from any cause), whichever came first, assessed at a minimum of 12 months.
  Measured using Response Assessment for Neuro-Oncology (RANO) criteria at screening, weeks 10, 22, 30 then 3 monthly (as per standard of care) for up to a minimum of 52 weeks from the start of trial treatment. PFS includes radiological progression assessed in accordance with RANO criteria and clinical progression where radiological progression is not possible.
Health-related quality of life (HRQoL) as assessed by EORTC QLQ-C30 | Baseline (Week 0), Week 8, Week 16, End of Treatment (Week 24)
  Generic Health-related quality of life (HRQoL) will be assessed with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) consisting of function, symptom and global health status scales, scored 1-4 with lower scores indicating better outcomes..
Adverse events | Baseline (Week 0), Week 4, Week 8, Week 12, Week 16, Week 20, End of Treatment (Week 24)
  Assessment of AEs according to the current NCI-CTCAE v5.0 criteria. Acute AE will be defined as those occurring up to 12 weeks post-end of treatment. Late AE will be defined as those occurring after 12 weeks post-end of treatment. The end of treatment will be the date of the final chemotherapy cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Collinson, MBBS, BSc, MRCP, FRCR, PhD, Principal Investigator — University of Leeds
Locations (22):
- United Kingdom (22):
  - Glan Clwyd Hospital, Bodelwyddan, Denbighshire
  - Mount Vernon Hospital, The Hillingdon Hospitals NHS Foundation Trust, Northwood, Middlesex
  - Aberdeen Royal Infirmary, NHS Grampian, Aberdeen
  - Belfast City Hospital, Belfast Health and Social Care Trust, Belfast
  - Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Bristol Haematology & Oncology Centre, University Hospitals Bristol & Weston NHS Foundation Trust, Bristol
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre Cancer Centre, Velindre University NHS Trust, Cardiff
  - Western General Hospital, NHS Lothian, Edinburgh
  - Beatson West of Scotland Cancer Centre, NHS Greater Glasgow & Clyde, Glasgow
  - Castle Hill Hospital, Hull University Teaching Hospitals NHS Trust, Hull
  - St James's University Hospital, Leeds Teaching Hospitals NHS Trust, Leeds
  - St Bartholomew's Hospital, Barts Health NHS Trust, London
  - Guy's Hospital, Guy's and St Thomas' NHS Foundation Trust, London
  - Charing Cross Hospital, Imperial College Healthcare NHS Trust, London
  - Maidstone Hospital, Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - The Christie Hospital, The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre, The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - City Hospital, Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Derriford Hospital, University Hospitals Plymouth NHS Trust, Plymouth
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Scientifically sound proposals from appropriately qualified researchers will be considered for data sharing. Requests should be made by returning a Data Sharing Request Form to newbusiness@trials.bham.ac.uk; this captures the research requirements, statistical analysis plan, and intended publication schedule. Requests will be reviewed by the Cancer Research UK Clinical Trials Unit (CRCTU) Directors in discussion with the Chief Investigator (CI), Trial Management Group (TMG) and independent Trial Steering Committee (TSC). They will consider the scientific validity of the request, qualifications of the researchers, views of CI, TMG and TSC, consent arrangements, practicality of anonymizing the requested data contractual obligations. If supportive of the request, and where not already obtained, Sponsor consent for data transfer will be sought before notifying applicants of the outcome. It is anticipated that applicants will be notified within 3 months of receipt of the original request.
Supporting Information: Study Protocol
URL: https://www.birmingham.ac.uk/research/centres-institutes/cancer-research-uk-clinical-trials-unit/data-sharing-policy

REFERENCES:
- [Background] Bhaskaran D, Savage J, Patel A, Collinson F, Mant R, Boele F, Brazil L, Meade S, Buckle P, Lax S, Billingham L, Short SC. A randomised phase II trial of temozolomide with or without cannabinoids in patients with recurrent glioblastoma (ARISTOCRAT): protocol for a multi-centre, double-blind, placebo-controlled trial. BMC Cancer. 2024 Jan 15;24(1):83. doi: 10.1186/s12885-023-11792-4. PMID 38225549
- See also: Trial Website — https://www.birmingham.ac.uk/aristocrat